CLINICAL TRIAL: NCT03769441
Title: Effect of Ferric Carboxymaltose on Exercise Capacity After Kidney Transplantation: a Multicenter Randomized Controlled Trial
Brief Title: Effect of Ferric Carboxymaltose on Exercise Capacity After Kidney Transplantation
Acronym: EFFECT-KTx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Kidney Foundation (Other); Vifor Fresenius Medical Care Renal Pharma (Industry)
Responsible Party: Principal Investigator, Martin H. de Borst, Principal Investigator, Clinical Professor, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201800450
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Iron-deficiency; Transplant-Related Disorder
Keywords: Renal Transplantation; Kidney Transplantation; Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is designed as a 24 week, multicentre, randomized placebo-controlled clinical trial with two parallel arms to investigate the effect of ferric(III) carboxymaltose on exercise tolerance, cardiac function, skeletal muscle function, quality of life, the gut microbiota and on the immune system, to be performed at the University Medical Center Groningen (UMCG) and the Erasmus MC, University Medical Center Rotterdam.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, care providers and researchers will be blinded, except for the nurse who will administer the medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric(III) carboxymaltose (Active Comparator): The intervention group will be treated with four dosages of 500 mg iron in the form of 10 mL ferric(III) carboxymaltose dissolved in 240 mL of NaCl 0.9%, with interval periods of six weeks.
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): The placebo-controlled group will receive four dosages of 250 mL of NaCl 0.9% solution with interval periods of six weeks.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Ferric carboxymaltose — Four intravenous dosages of ferric(III) carboxymaltose
  Arms: Ferric(III) carboxymaltose
Drug: Sodium chloride — Four intravenous dosages of sodiumchloride
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Iron deficiency is common in kidney transplant recipients and is associated with impaired exercise tolerance and an unfavourable prognosis.

This multicentre double-blind, placebo-controlled randomized controlled clinical trial will allow the investigators to analyse the effects of intravenous iron correction with ferric(III) carboxymaltose on exercise tolerance and other parameters, in comparison to a placebo.

DETAILED DESCRIPTION:
Rationale: Iron deficiency is common in kidney transplant recipients. The presence of iron deficiency is associated with an unfavourable prognosis in these patients. In patients with heart failure and iron deficiency, treatment with intravenous iron improved exercise capacity and quality of life. Whether such beneficial effects may also occur in kidney transplant recipients is unknown.

Objective: Our main objective is to address whether correction of iron deficiency with ferric(III) carboxymaltose improves exercise tolerance and quality of life in iron-deficient kidney-transplant recipients.

Study design: A multicentre double-blind, placebo-controlled randomized controlled clinical trial will be performed to compare the effects of ferric(III) carboxymaltose with placebo.

Study population: 158 iron-deficient kidney transplant recipients. The intervention arm will receive 10 mL of ferric(III) carboxymaltose (50 mg Fe3/mL, intravenously) every six weeks, with a total of four dosages. The control arm receives an intravenous placebo solution (saline).

Main study parameters/endpoints: The primary endpoint is the distance walked in six minutes, as quantified by the six-minute-walking-test at the end of follow-up.

The investigators expect that iron-deficient kidney transplant recipients will benefit from ferric(III) carboxymaltose treatment as a result of an improvement in exercise tolerance and general wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient
* Iron deficiency, defined by a ferritin level of ≤100 ug/L, or 100-299 ug/L combined with a transferrin saturation of ≤20%
* At least six months after transplantation at baseline
* Age ≥18 years
* Ability to comply with the study protocol
* Informed consent

Exclusion Criteria:

* Intolerance to any intravenous iron solution
* Severe anemia (Hb <10.5 g/dL, <6.5 mmol/L), microcytic anemia (MCV <80 fl) or progressive anemia (˃3.2 g/dL per month decline for two months or more)
* A positive feces occult blood test or otherwise demonstrated gastrointestinal, or urogenital, blood loss
* Blood transfusion in the past six weeks
* Polycythemia (Hb >15.3 g/dL, 9.5 mmol/L)
* Estimated glomerular filtration rate (eGFR) of ≤ 30 ml/min per 1.73 m2
* History of haemochromatosis
* Unstable angina or myocardial infarction during the previous month
* Disability to walk
* Severe hypophosphatemia in the month before baseline (serum phosphate <0.35 mmol/L)
* Pregnancy or inability to take adequate contraceptive measures when at childbearing age (women)
* Any signs of an active systemic infection
* Participation in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | 24 weeks
  The between-group difference in change in exercise tolerance quantified by the six-minute walk test (6MWT)

SECONDARY OUTCOMES:
Hemoglobin level | 24 weeks
  The between-group difference in change in hemoglobin level
Iron status | 24 weeks
  The between-group difference in change in iron parameters (plasma iron, ferritin, transferrin saturation)
Cardiac function | 24 weeks
  The between-group difference in change in cardiac structure, function and strain, analysed with a transthoracic echocardiography
Muscle strength 1 | 24 weeks
  The between-group difference in change in muscle strength measured by the 'Five-Times-Sit-to-Stand-test (FTSTS)
Muscle strength 2 | 24 weeks
  The between-group difference in change in muscle strength measured by the timed-up-and-Go test (TUG)
Muscle strength 3 | 24 weeks
  The between-group difference in change in muscle strength measured by handgrip dynamometry
Muscle mass | 24 weeks
  The between-group difference in change in muscle mass assessed using 24-hour urinary creatinine excretion
Phosphate level | 24 weeks
  The between-group difference in change in phosphate level
Calcium level | 24 weeks
  The between-group difference in change in calcium level
Vitamin D status | 24 weeks
  The between-group difference in change in vitamin D level
Parathyroid hormone | 24 weeks
  The between-group difference in change in parathyroid hormone level level
FGF23 | 24 weeks
  The between-group difference in change in FGF23 level
Intestinal microbiota | 24 weeks
  The between-group difference in change in intestinal microbiota
Incidence of any infection | 24 weeks
  The between-group difference in incidence of infections
Incidence of hospitalisation | 24 weeks
  The between-group difference in incidence of hospitalisation
Incidence of cardiac events | 24 weeks
  The between-group difference in incidence of cardiac events
Incidence of graft failure | 24 weeks
  The between-group difference in incidence of graft failure
Lymphocyte production of cytokines | 24 weeks
  The between-group difference in lymphocyte cytokine espression (measured with facs)
Lymphocyte production of immunoglobulins | 24 weeks
  The between-group difference in lymphocyte IgG production (measured with ELISA)
Lymphocyte proliferation rate | 24 weeks
  The between-group difference in lymphocyte proliferation rate (assessed with FACS)
B-lymphocyte differentiation rate | 24 weeks
  The between-group difference in B-lymphocyte plasma cell formation (assessed with Facs)
Cognitive performance (memory span) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (Digit Span Forward Test, minimum value 0, maximum value 9, a higher score means a better outcome)
Cognitive performance (verbal memory) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (15 word test, minimum value 0, maximum value 75, a higher score means a better outcome)
Cognitive performance (semantic memory) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (Word Fluency Test, minimum value 0, no maximum value, a higher score means a better outcome)
Cognitive performance (processing speed) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (symbol digit modalities test, minimum value 0, maximum value 110, a higher score means a better outcome)
Cognitive performance (visuomotor and mental speed) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (Trail Making Test A, minimum value 1, no maximum value, a lower score means a better outcome)
Cognitive performance (cognitive flexibility) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (Trail Making Test B, minimum value 1, no maximum value, a lower score means a better outcome)
Cognitive performance (executive control) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (Controlled Oral Word Association Test, minimum score 1, no maximum score, a higher score means a better outcome)
Cognitive performance (working memory) | 24 weeks
  The between-group difference in change in cognitive performance quantified with neuropsychological testing (Digit Span Backward, minimum score 0, maximum score 8, a higher score means a better outcome)
Plasma creatinine | 24 weeks
  The between-group difference in change in plasma creatinine
Quality of Life (health) | 24 weeks
  The between-group difference in change in quality of life quantified with SF36 questionnaire. A higher score means a better outcome.
Quality of Life (subjective fatigue) | 24 weeks
  The between-group difference in change in quality of life quantified with the Dutch Checklist individual Strength). A higher score means worse fatigue.
Quality of Life (long-lasting fatigue) | 24 weeks
  The between-group difference in change in quality of life quantified with the Dutch Multifactor Fatigue Scale). A higher score means worse fatigue.
Quality of Life (overall) | 24 weeks
  The between-group difference in change in quality of life quantified with EuroQol-5D-5L
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccination IgG response | 12 months
  The between-group difference in severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) specific antibody titre after vaccination.
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccination T-lymphocyte response | 12 months
  The between-group difference in severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) specif T-lymphocyte response after vaccination.
Gastro-intestinal symptoms | 24 weeks
  The between-group difference in change in gastro-intestinal symptoms assessed with the gastrointestinal symptom rating scale.
Hepatic injury | 24 weeks
  The between-group difference in change in plasma hepatic enzyme levels (aspartate transaminase and alanine transaminase)
Restless legs | 24 weeks
  The between-group difference in prevalence of restless legs symptoms before and after treatment
Kidney graft rejection and injury | 24 weeks
  The between-group difference in change in urine kidney injury marker levels

CONTACTS AND LOCATIONS:
Overall Officials: Martin de Borst, MD/PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
To protect participant privacy, public access to the dataset or individual participant data will not be provided. However, after deidentification of these data and after publication of the main results, requests for the re-use of all pseudo-anonymised individual participant data by researchers who provide a methodologically sound proposal for a secondary analysis or meta-analysis will be evaluated by the Principal Investigator. Data may be shared if the research question falls within the scope of the informed consent. Proposals should be directed to m.h.de.borst@umcg.nl and requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol, including a statistical data analysis plan, will be published in a peer-reviewed journal.

REFERENCES:
- [Derived] Vinke JS, Eisenga MF, Sanders JF, Berger SP, Spikman JM, Abdulahad WH, Bakker SJ, Gaillard CAJM, van Zuilen AD, van der Meer P, de Borst MH. Effect of Intravenous Ferric Carboxymaltose on Exercise Capacity After Kidney Transplantation (EFFECT-KTx): rationale and study protocol for a double-blind, randomised, placebo-controlled trial. BMJ Open. 2023 Mar 22;13(3):e065423. doi: 10.1136/bmjopen-2022-065423. PMID 36948568